CLINICAL TRIAL: NCT00733668
Title: An Open-Label, Non-Comparative, Multi-Centre, Phase II Prospective Trial to Assess the Efficacy of Quetiapine Fumarate Augmentation of Selective Serotonin Reuptake Inhibitors (SSRIs) in SSRI-Resistant Major Depressive Disorder.
Brief Title: Efficacy of SEROQUEL in Selective Serotonin Reuptake Inhibitors (SSRI)-Resistant Major Depressive Disorder
Acronym: UNIQUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: An Matthys, MD, Therapeutic Area Leader CNS, AstraZeneca Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1449C00009
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Major Depressive Disorder
Keywords: considered; entry; into; the study; SSRI; Seroquel; Quetiapine; fumarate; antipsychotic
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Quetiapine fumarate (Seroquel) — 300 mg, PO, 100 mg morning, 200 mg evening, 4 weeks
  Other Names: Seroquel

SUMMARY:
An open-label, non-comparative, multi-centre, phase II prospective trial to assess the efficacy of Quetiapine fumarate augmentation of selective serotonin reuptake inhibitors (SSRIs) in SSRI-resistant major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Inform consent
* Male and female, age between 18 and 65 years.
* Naïve to any atypical antipsychotic
* A diagnosis of major depressive disorder

Exclusion Criteria:

* No use of fluvoxamine
* Patients with a history of bipolar I or II disorder
* Diagnosis of psychotic major depression disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The Montgomery-Asberg Depression Scale (MADRS) score | Visit 1 - > 5

SECONDARY OUTCOMES:
The Brief psychiatric Rating Scale (BPRS) scoreThe Clinical Global impression (CGI) scorePatient reported outcomes (PROs) | Visit 1 - > 5 (1 week between each visit)
Sheehan Disability Scale (SDS) score | Visit 1 - > 5 (1 week between each visit)
The Symptom Checklist 90 Revisred (SCL-90-R) score | Visit 1 - > 5 (1 week between each visit)

CONTACTS AND LOCATIONS:
Overall Officials: Pr. Demyttenaere, Study Director — KUL
Locations (4):
- Belgium (4):
  - Research Site, Bruges
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Sint-Truiden